CLINICAL TRIAL: NCT05619237
Title: Act to Improve Chronic Wounds in Alberta: Pivotal Study on the Use of NanoSALV Antimicrobial Wound Dressing to Treat Chronic Wounds
Brief Title: Pivotal Study of an Antimicrobial Wound Dressing to Treat Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chester Ho, MD (Other)
Collaborators: Alberta Health services (Other); NanoTess Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Chester Ho, MD, Spinal Cord Injury Research Chair and, University of Calgary
Organization: University of Calgary (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB22-1394
Record Dates: First submitted 2022-11-02; First posted 2022-11-16 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pressure Injury; Venous Leg Ulcer; Pressure Injury Stage 2; Pressure Injury Stage III; Diabetic Foot Ulcer; Pressure Injury Stage IV; Leg Ulcer
Keywords: pressure injury; chronic wound
MeSH Terms: conditions — Pressure Ulcer; Varicose Ulcer; Diabetic Foot; Leg Ulcer

STUDY DESIGN:
Intervention Model Description: Patients will receive the standard of care for the first 4 weeks. If the chronic wound has healed less than 50%, then the patient will receive the intervention for 4 weeks.
Masking Description: Participants and researchers will be aware of the phases of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Period (No Intervention): Patients receive the current standard of care for their chronic wound in the first four weeks of enrollment
  Standard of care (SOC) involves:
  * Offloading of pressure as needed
  * High compression bandaging, as needed
  * Debridement, as needed
  * Nutrition management, as needed
  * SOC dressings, such as silver/iodine dressings, antibiotic ointment
  * Management of infection
  * Management of pain during debridement, as needed
- Intervention Period (Experimental): Patients receive the intervention, NanoSALV wound dressing, in the consecutive four weeks following the control period
  Interventions: Device: NanoSALV Catalytic

INTERVENTIONS:
Device: NanoSALV Catalytic — NanoSALV Catalytic Antimicrobial Wound Dressing Gel is a Health Canada approved medical device for the management of Chronic Wounds.
  Arms: Intervention Period

SUMMARY:
The goal of this clinical trial is to assess the impact that the NanoSALV wound dressing can have on managing severe chronic wounds and feasibility for patients, providers, and health systems in different health care settings (community care, continuing care and in-patient care).

The main questions it aims to answer are:

1. What is the cost-savings of using NanoSALV?
2. Do care providers perceive NanoSALV to be better, worse or the same as the standard of care in terms of usability and efficiency?
3. Does NanoSALV increase autonomy and competence of wound self-management for care providers/patients?
4. Were patients more satisfied, less satisfied or just as satisfied with NanoSALV compared to the standard of Care?
5. Does NanoSALV reduce healing time for chronic wounds compared to standard of care?

The sequence and duration of the trial is as follows:

* Required data will be collected at enrollment to provide a baseline (Day 0) measure.
* The patient will receive standard of care treatment for four weeks with dressing changes as per the standard care pathway.
* In the following four weeks the patient will receive the NanoSALV dressing treatment and dressing changes done every 48 - 72 hours as required.
* Wound assessments will be done weekly with wound images captured by Aranz Medical's Silhouette Star 3D medical camera that digitally takes measurements.
* A patient satisfaction survey will be collected post-control and post-intervention periods
* One week after completing the study the patient/surrogate will be contacted or a survey link will be sent to them regarding adverse events and to see what wound dressing they continued to use.

Semi-structured interviews and observations will be done with care providers/patients and healthcare professionals in the control period to explore the perspectives on the current state of chronic wound management, and in the intervention period to evaluate the perceptions on the usability of the intervention.

DETAILED DESCRIPTION:
1. BACKGROUND:

   Chronic wounds include, but are not limited, to diabetic foot ulcers (DFU), venous leg ulcers (VLU), and pressure ulcers. They are a challenge to wound care professionals and consume a great deal of healthcare resources. Chronic wounds are defined as wounds that fail to proceed through the normal phases of wound healing in an orderly and timely manner. Venous Leg Ulcer (VLU) is a recurrent chronic wound on the lower leg, and it is associated with venous obstruction or reflux, both of which also lead to poor venous flow and venous hypertension. A pressure injury (also known as a pressure ulcer) is defined by the National Pressure Injury Advisory Panel as a "localized damage to the skin and underlying soft tissue usually over a bony prominence or related to medical or other devices. The injury can present as intact skin or an open ulcer and may be painful". The development of a pressure injury is influenced by a variety of factors including age, mobility, nutrition, and other comorbid diseases/conditions. DFU is a frequent complication and hospitalization for individuals with diabetes mellitus (DM). As a result, these regions with limited sensitivity and chronic trauma can progress to an ulcer, potentially causing ischemia to the deep tissues, sometimes including the bone. These ulcerative tissues are highly susceptible to colonization and infection by multiple bacteria, and often result from the improper lack of care (debridement, antibacterials, etc). More severe DFUs may require surgical intervention and amputation, to prevent progression.

   Pressure injuries have significant negative consequences for both patients and the health system. They compromise patient health outcomes, have been found to cause pain, hinder functional recovery and present a high risk for the development of serious infections. They have also been associated with an extended length of stay, sepsis and mortality. In a similar manner, VLU has significant social and economic burden to the patient and the healthcare system. Patient mobility, health-related quality of life, social roles, employment, and physical activity are negatively affected by this condition. Furthermore, besides the high quality of life and mortality burden related to DFU and amputations, health care costs and economic burden related to this issue are also high. Patients with DM complications, such as DFU, require frequent and significant medical care with expensive medical supplies and are often unable to work due to disease management issues and disability/mobility challenges.

   Currently, the most effective practices for the treatment of chronic wounds involve: Cleansing (e.g.: with sterile water or saline), Debriding (e.g.: autolytic, mechanical, enzymatic etc.), managing bacterial balance (e.g.: with antibiotics) and managing moisture balance (e.g.: with draining). Dressings are recommended to promote healing (e.g.: to support drainage and provide tissue protection) and prevent infection (e.g.: antimicrobial products such as those impregnated with silver, honey or iodine). However, these products have drawbacks such as: not being able to conform to or sufficiently cover the wound, pain with wearing and/or removal, and only functioning to either promote healing OR treat the infection. An innovative solution should have features such as the ability to conform to the wound regardless of wound topography, be able to be worn for long periods, not be painful to wear, and have combined actions to simultaneously promote healing and be antimicrobial.

   NanoSALV is a hydrogel wound dressing that contains NanoKARE technology, which is an advanced composite material that provides broad-spectrum antimicrobial and catalytic effects that reduce the thresholds needed to achieve optimal healing potential. NanoSALV wound dressing gel provides broad-spectrum antimicrobial effect against bacteria, fungi and viruses, and catalytic effects to achieve optimal healing potential. Has passed skin sensitization, irritation, acute systemic toxicity, and cytotoxicity during in-vitro testing. There are no known adverse events or reactions.

   Antimicrobial efficacy in-vitro testing of NanoKARE technology ranged from 0.5-6% for minimum inhibitory concentration (MIC) and 0.5-8% minimum bactericidal concentration (MBC) for all microorganisms tested. MIC/MBC testing was performed by JMI Laboratories. Biofilm in-vitro testing showed the technology was effective at eliminating all resistant biofilms tested and effectively prevented the formation of all biofilm strains. SARS-CoV-2 in-vitro surface testing also showed 99.9% reduction in viral strains after 30s of exposure and lasted up to 7 days after a single surface application. These tests were fully funded by the Canadian Department of Defense.
2. OBJECTIVE:

   Objective: To assess the implementation feasibility and impact that a potential innovative solution NanoSalv to manage severe chronic wounds and pressure injuries may bring to the patient, provider and health system.
3. METHODS:

Patients with diabetic foot ulcers, venous leg ulcers and stage II to IV pressure injuries will be recruited. Each patient will receive four weeks of the standard of care and four weeks of the intervention.

Weekly wound assessments will be done and wound images will be captured by a 3D medical camera that digitally takes measurements. Patients will be shown their wound images to show their progress of wound healing.

To explore the perspectives on the current state of chronic wound management, review of care plan protocols, policies and procedures, Likert scales, and semi-structured interviews and observations will be done with care providers/patients and healthcare professionals from the different sites during the control period. To evaluate the perceptions on the usability of and experience with the intervention, semi-structured interviews and observations, and Likert scales will be done with the previously mentioned users of the intervention in the intervention period throughout the project implementation. The data collected will be analyzed using journey mapping, comparative task analysis, thematic analysis, and workflow analysis.

Sample Size:

The sample size was determined based in part on the feasibility of recruiting patients in the given timeline and the project personnel provided. A sample size of 95 patients with 10 weeks to recruit would average recruiting 8-9 patients per week. For the qualitative methods involving semi-structured interviews on current perspectives of standard care, interviews on perceptions, and usability of the intervention, 9-20 participants will be recruited to participate over the duration of the study period.

The sequence and duration of all trial periods is as follows:

Initiation:

* Potential participants will be identified by healthcare providers
* Research Staff will screen for eligibility with the Principal Investigator/Co-Investigator or the patient's attending physician and will consent eligible patients
* Required data will be collected about the patient and the wound at enrollment to provide a baseline measure on Day 0: Patient demographics (age, sex, type of wound), Charlson Comorbidities, wound measurements area and volume and photographs (using a 3D wound camera), and wound assessments (e.g., Bates-Jensen Wound Assessment Tool (BWAT), infection, pain)
* The wound will be debrided and cleaned as required by wound care

Control Period:

* The patient will receive standard of care treatment for 4 weeks with dressing changes as per the standard care pathway.
* Wound measurements, images and assessments will be done every 7 days for weekly data collection
* Data collected on Day 7, 14, 21: wound area, volume, assessments and photographs (e.g., BWAT, infection, pain), dressing and standard of care (SOC) compliance
* On day 28 all patient wounds will be evaluated for the inclusion criteria: percentage area reduction of the wound ≤ 50%.
* Data collected on Day 28: wound area, volume assessments and photographs (e.g., BWAT, infection, pain), dressing compliance, patient satisfaction
* Wound clinic staff, long-term care (LTC) staff and patient/family caregivers will be asked to participate in 1h semi-structured interviews

Intervention Period:

* Day 29, patient will start using the NanoSALV intervention and dressing changes done every 48 - 72 hours as required.
* Patient and wound will be assessed every 7 days for weekly data collection
* Data collected on Day 35, 42 and 49: wound area and volume assessments and photographs (e.g., BWAT, infection, pain), dressing compliance
* Data collected on Day 56: wound area and volume assessments and photographs (e.g., BWAT, infection, pain), wound QoL-14 (Note for wound clinic patients this will be done at the clinic), dressing compliance, patient satisfaction
* Wound clinic staff, LTC staff and patient/family caregivers will be asked to participate in 1h semi-structured interviews

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years or over
* Provide informed consent or have a legal representative consent on their behalf
* Ability and willingness to adhere to the study requirements including weekly appointments and required site visits.
* Ability and willingness to comply with standard of care practices as per the type of wound
* Suspect chronic wound being treated with standard of care for at least 14 days

Chronic wound inclusion criteria:

Pressure Injury

* Stage II, III, or IV
* Ulcer area post debridement between 2cm^2 and 50cm^2

Diabetic Foot Ulcer

* Have a diagnosis of diabetes mellitus type 1 or 2 or pre-diabetic
* Ulcer area post debridement between 1cm^2 and 25cm^2

Venous / Leg Ulcer

- Ulcer area post debridement between 2cm^2 and 50cm^2

Exclusion Criteria:

* Life expectancy less than 6 months
* Not responding to treatment for osteomyelitis and/or sepsis
* Presence of necrotic debris and/or gangrene post debridement is greater than 75% of wound surface area
* Fall within the contraindications of the intervention product (allergies to the any of the ingredients, pregnant or breast feeding)
* Currently participating in another study that would interfere with this study or would overburden the patient if enrolled in this study
* Presence of a life-threatening disease with no current treatment plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Soft Cost Savings | Through study completion over four months
  Evaluation of the cost savings during the intervention period compared to the control period, by tracking indirect and direct costs including but not limited to, wound dressing costs, duration of treatment, frequency of dressing changes, in-clinic visit frequency, time and duration, in-home patient care, wound reduction rates, expenditure during control period and expenditure during intervention period, etc. This would be evaluated by a health economist and economic analysis support by the study sponsor.
User Satisfaction | Through study completion over four months
  Qualitative evaluation of the patient's and care provider's satisfaction with the Innovation in comparison to standard of care to inform future adoption decisions.
  Measured by: follow-up with User's desire to continue intervention over standard of care wound dressings as measured by the number of user's who sign up to continue with the intervention.
User Experience | Through study completion over four months
  Qualitative evaluation of the patient's and care provider's experience with the Innovation in comparison to standard of care to inform future adoption decisions.
  Measured by: Semi-structured interview themes will also be recorded to understand enablers and barriers to product use.
Process Improvement | Through study completion over four months
  Evaluation of workflow considerations with the Innovation in comparison to the standard of care.
  Measured by: documenting the frequency of dressing changes, and person who completes dressing changes to determine adoption and ability to change dressings outside of a healthcare setting. Task analysis will be conducted during the control and intervention to compare differences and similarities in tasks required to change dressing.
Quality Improvement | Through study completion over four months
  Evaluation of performance with the Innovation in comparison to the standard of care.
  Measured by: Subjective observations by human factors study team will be documented and follow-up interviews will be coded to reflect themes of enablers and barriers to standard of care vs intervention

SECONDARY OUTCOMES:
Wound percent area change | Weekly assessments over 8 weeks
  Measured by: photographs of the wound using Aranz Silhouette Star 3D camera followed by wound area tracing and area analysis using Aranz Silhouette Star software.
Wound percent volume change | Weekly assessments over 8 weeks
  Measured by: photographs of the wound using Aranz Silhouette Star 3D camera followed by wound area tracing and volume analysis using Aranz Silhouette Star software.
Adverse events | Through study completion over four months
  Measured by: the number of confirmed adverse events documented.
Patient preference | Weekly assessments over 8 weeks
  Evaluation of the patient's satisfaction with the use of NanoSALV in comparison to standard of care.
  Measured by: Patient's choice of continuing with SOC or NanoSALV after study completion
Patient satisfaction - ease of use | Change between Day 28 and Day 56 of study enrollment
  Evaluation of the patient's satisfaction with the use of NanoSALV in comparison to standard of care.
  Measured by: comparing patient satisfaction surveys post control and intervention periods using 10-point Likert scales assessing ease of use
Patient satisfaction - comfort | Change between Day 28 and Day 56 of study enrollment
  Evaluation of the patient's satisfaction with the use of NanoSALV in comparison to standard of care.
  Measured by: comparing patient satisfaction surveys post control and intervention periods using 10-point Likert scales assessing comfort of wound dressing
Patient satisfaction - overall satisfaction | Change between Day 28 and Day 56 of study enrollment
  Evaluation of the patient's satisfaction with the use of NanoSALV in comparison to standard of care.
  Measured by: comparing patient satisfaction surveys post control and intervention periods using 10-point Likert scales assessing overall satisfaction with wound dressing

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Carewest Dr. Vernon Fanning Long-Term Care, Calgary, Alberta
  - Sheldon Chumir Wound Clinic, Calgary, Alberta
  - Calgary Foot Care Nurses Clinic, Calgary, Alberta
  - Glenrose Rehabilitation Centre, Edmonton, Alberta